CLINICAL TRIAL: NCT05302180
Title: Online Pain Education in Addition to Usual Care in Individuals With Chronic Musculoskeletal Pain: Protocol for a Hybrid Type III Randomized Controlled Trial.
Brief Title: Online Pain Education in Addition to Usual Care in Chronic Pain.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Cidade de Sao Paulo (Other)
Responsible Party: Principal Investigator, Dr Bruno Saragiotto, Clinical professor, Universidade Cidade de Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 11975019.0.0000.0106
Record Dates: First submitted 2022-02-15; First posted 2022-03-31 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Chronic Pain; Musculoskeletal Pain
MeSH Terms: conditions — Chronic Pain; Musculoskeletal Pain

STUDY DESIGN:
Intervention Model Description: hybrid type III effectiveness-implementation randomized controlled trial
Who Masked: Investigator
Masking Description: The outcomes' evaluators will be blind about the allocation of participants in the study groups and they will be questioned at the end of the study on which group they believe that each participant was allocated in order to evaluate the success/failure of blinding. Due to the nature of the interventions it will not be possible to blind the participants and researchers responsible for the interventions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Synchronous online group (Experimental): The synchronous online pain neuroscience education program (EducaDor program) will be held in groups at until 12 participants, at 10 weekly synchronous meetings on the Whereby® platform.The professional will conduct each synchronous meeting with dialogued exhibition class using multimedia material shared on the computer screen
  Interventions: Other: Pain neuroscience education; Other: Usual care
- Asynchronous group (Experimental): Participants allocated in the asynchronous group will receive the interactive e-book at the beginning of the program and ten videos (one per week) with the same topics of synchronous online EducaDor program sent on their smartphone devices and e-mail, in addition to usual care. Before receiving the materials, users will participate in an individual or group synchronous meeting of up to 12 participants on the Whereby® platform to receive a guidance for the use of interactive e-book and access to videos over the 10 weeks. The videos were previously developed and tested in another clinical trial.
  Interventions: Other: Pain neuroscience education; Other: Usual care
- E-book group (Active Comparator): Participants allocated to this group will receive the interactive e-book of EducaDor program in their smartphone devices and e-mail, in addition to usual care. Before receiving the e-book, the users will also participate in an individual or group synchronous meeting of up to 12 participants on the Whereby® platform to receive a guidance for the use of interactive e-book over the 10 weeks.
  Interventions: Other: Pain neuroscience education; Other: Usual care

INTERVENTIONS:
Other: Pain neuroscience education — The online pain neuroscience education program will be based on the model proposed by the Pain Research Group, available in http://pesquisaemdor.com.br, which presents the "Path of Recovery". In our program we will hold 10 meetings: (1) conversation with the group, (2) acceptance and pain education, (3) continuation about pain education, (4) sleep hygiene, (5) pharmacological assistance, (6) recognizing stress and negative emotions, (7) increasing positive coping in lifestyle, (8) exercises, (9) communication, and (10) prevention of recurrence. The program will be offered by synchronous meetings; asynchronous (videos) and e-book.
Other: Usual care — All participants will receive usual care in one of the five physiotherapy clinics accredited to SUS, according to availability of scheduling in the services. The usual care consists of 10 sessions of physical therapy, that is mainly composed by kinesiotherapy and electrothermophototherapy.

SUMMARY:
The lack of pain specialists limits users' access to non-pharmacological therapeutic pain control strategies. In this context, digital health programs can reduce the inequity of access to interventions, contribute to the self-management of chronic musculoskeletal conditions, reduce the burden on primary care and can help to reorganize the flow of referral of individuals in the health care network. The aim of this study will be to analyze the implementation and health outcomes of three online pain neuroscience education strategies in individuals with chronic musculoskeletal pain. This is a hybrid type III effectiveness-implementation randomized controlled trial. Individuals with ≥18 years old with chronic musculoskeletal pain will be recruited from primary health care in the city of Guarapuava/PR/Brazil and referred to the health care network for conventional physical therapy in addition to the online pain neuroscience education program (EducaDor). The EducaDor program will be delivered in 3 modalities: 1) synchronous online; 2) asynchronous videos; 3) Interactive e-book. The implementation outcomes evaluated will be: acceptability, appropriateness, feasibility, adoption, fidelity, penetration, sustainability and costs; and health outcomes will include: pain, functionality, quality of life, sleep, physical activity, self-efficacy, adverse effects, prognostic and risk groups. The evaluations will be done at baseline, after the end of the interventions and follow-up of 6 months.

DETAILED DESCRIPTION:
Systematic reviews have demonstrated the efficacy of pain neuroscience education in the treatment of adult individuals with chronic musculoskeletal pain in reducing pain, anxiety, and depression; and increased of knowledge about pain, functionality and physical performance. The literature demonstrates moderate quality of evidence of pain neuroscience education in addition to usual physical therapy intervention in short-term with a weighted mean difference of 1.3 points for pain and 3.94 points for disability. Previous systematic reviews also suggest that pain neuroscience education alongside to usual physical therapy care or exercise-based treatments can be considered cost-effective compared to usual care alone.

Despite the large evidence for treatment of chronic pain, generally these evidence-based strategies are inadequately applied in practice by public health providers, inadequately integrated into lifestyle behaviors by health users and featured in health policy and health service delivery at a disproportionate level with the burden of disease. Another point, is that most of this available evidence is derived largely from research of high-income economies and reflected in clinical practice guidelines and policies targeted towards high-income settings. So, strategies to translate this evidence into policy and practice in low- and middle-income settings remain sparse. Hence, implementation research to determine the most acceptable, effective and sustainable health strategies to bring the chronic pain clinical practice guidelines into policy and practice in low- and middle-income countries is urgently needed.

Thus, the implementation of an online pain neuroscience education service in the health care network of Brazilian Unified Health System (SUS) articulated with primary health care could provide coordinated and consistent care to the needs of individuals with chronic pain, with appropriate reference to specialists. The purpose of this study is to conduct a hybrid type III effectiveness-implementation randomized controlled trial with the following objectives: (1) to assess the effects of three implementation strategies of an online pain neuroscience education service in the public health system of Guarapuava city, Parana, Brazil; (2) to compare the effectiveness and cost-effectiveness of the three implementation strategies of online pain education.

ELIGIBILITY:
Inclusion Criteria:

1. individuals that report musculoskeletal pain in the last 3 months;
2. can read and write in Portuguese language;
3. have smartphone, tablet or computer with internet access.
4. Participants will be included in the study after agreeing and signing the Informed Consent Form (ICF).

Exclusion Criteria:

There will be no exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 249 (Estimated)
Dates: Start 2022-10-27 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Change from baseline pain at 10 week of the intervention | baseline, 10 week
  numerical rating scale (NRS) of 11 points, ranging from 0 (no pain) to 10 points (the worst possible pain) points
Maintenance of pain at 6 months of the intervention | up to 6 months
  numerical rating scale (NRS) of 11 points, ranging from 0 (no pain) to 10 points (the worst possible pain) points

SECONDARY OUTCOMES:
Change from baseline self-efficacy at 10 week of the intervention | baseline, 10 week
  Chronic Pain Self-Efficacy Scale (CPSS)(63), with 22 items of individual's beliefs, whose items are divided into three factors: (1) self-efficacy for pain control (AED), (2) self-efficacy for other symptoms (AES) and (3) self-efficacy for physical function (AEF). It is possible to obtain a score for each factor (score ranging from 10 to 100), and the sum of all factors that ranges from 30 to 300 points
Change from baseline function at 10 week of the intervention | baseline, 10 week
  The Patient Specific Functional Scale (PSFS-Br) will be used. The participant appoint 3 to 5 important activities which they have greater difficulty due to their condition and then graduates the level of their difficulty on a 11 points scale, ranging 0 (inability to perform the activity) to 10 (capable of performing the activity at the same level as before the injury or problem)
Maintenance of function at 6 months of the intervention | up to 6 months
  The Patient Specific Functional Scale (PSFS-Br) will be used. The participant appoint 3 to 5 important activities which they have greater difficulty due to their condition and then graduates the level of their difficulty on a 11 points scale, ranging 0 (inability to perform the activity) to 10 (capable of performing the activity at the same level as before the injury or problem)
Change from baseline quality of sleep at 10 week of the intervention | baseline, 10 week
  Quality of sleep will be evaluated by a self-report of sleep quality in the last 7 days on a scale of 0 to 100 points (0 - worst sleep quality; 100 - better sleep quality).
Maintenance of quality of sleep at 6 months of the intervention | up to 6 months
  Quality of sleep will be evaluated by a self-report of sleep quality in the last 7 days on a scale of 0 to 100 points (0 - worst sleep quality; 100 - better sleep quality).
Change from baseline physical activity at 10 week of the intervention | baseline, 10 week
  Physical activity will be evaluated by a self-report of the type, duration and intensity of physical activity performed in the last 7 days
Maintenance of physical activity at 6 months of the intervention | up to 6 months
  Physical activity will be evaluated by a self-report of the type, duration and intensity of physical activity performed in the last 7 days
Change from baseline health-related quality of life at 10 week of the intervention | baseline, 10 week
  Health-related quality of life: will be evaluated using the EQ-5D-3L questionnaire, which is composed of a descriptive model with five health domains (mobility, self-care, usual activities, pain/discomfort, anxiety/depression).
Maintenance of health-related quality at 6 months of the intervention | up to 6 months
  Health-related quality of life: will be evaluated using the EQ-5D-3L questionnaire, which is composed of a descriptive model with five health domains (mobility, self-care, usual activities, pain/discomfort, anxiety/depression).
Change from baseline prognostic and risk groups at 10 week of the intervention | baseline, 10 week
  Prognostic and risk groups will be evaluated by the Keele STarT MSK Took(67). The tool contains 10 items (ranged from 0 to 12 points each) that once scored can place patients into three categories based on their risk of a poor outcome in low risk (0-4 points), medium risk (5-8 points), and high risk (9-12 points)
Maintenance of prognostic and risk groups at 6 months of the intervention | up to 6 months
  Prognostic and risk groups will be evaluated by the Keele STarT MSK Took(67). The tool contains 10 items (ranged from 0 to 12 points each) that once scored can place patients into three categories based on their risk of a poor outcome in low risk (0-4 points), medium risk (5-8 points), and high risk (9-12 points)
Occurrence of adverse events up to 6 months of the intervention begging | 10 week; and up to 6 months
  Adverse events: will be analyzed by recording the number and type of adverse effects that occurred during the intervention period.

OTHER OUTCOMES:
Assessment of the intervention acceptability by the perspective of public health managers | through study completion, an average 24 months
  will be analyzed from the perspective of public health managers through focus group interview, and the Acceptability of Intervention Measure (AIM) will be used.
Assessment of the intervention acceptability by the perspective of participants | 10 week
  will be analyzed from the perspective of participants by individual qualitative interview about satisfaction with the intervention and by a numerical scale from 0 to 100 of how satisfied they were with participation in the intervention. The Acceptability of intervention measure (AIM) will be used.
Assessment of the intervention appropriateness by the participants' perspective | 10 week
  Appropriateness will be analyzed from the participant's perspective regarding the perception of appropriateness of each component EducaDor program for their health condition through an adapted questionnaire used by Liao et al (2020). This questionnaire will assess the degree to which participants agree with a series of statements about the intervention, on a likert scale ranging from 1 (totally disagree) to 4 (totally agree). An individual qualitative interview ill also be conducted with EducaDor program's participants in order to identify the barriers and facilitators of the proposed interventions. The Intervention appropriateness measure (IAM) will also be used.
Assessment of the intervention feasibility by the organization and individual providers | through study completion, an average 24 months
  Feasibility will be evaluated from the perspective of the organization and individual providers through a focus group interview. The Feasibility intervention measure (FIM) will be used.
Assessment of the intervention adoption | pre-intervention
  Adoption will be analyzed by the percentage of acceptance of public health users to participate in EducaDor program referred from primary health care. Those public health users that refuse to participate, during telephone contact will be done an individual qualitative interview to identify barriers to engagement to EducaDor program.
Assessment of the intervention fidelity by perspective of the specialist | through study completion, an average 24 months
  Fidelity will be evaluated by an independent pain specialist, who will randomly select 10% of the recorded meetings and evaluate them in relation to the fidelity of the intervention manuals with the content and quality of the meetings in a qualitative individual interview.
Assessment of the intervention fidelity by the adherence of participants during 10 week intervention | 10 week
  The adherence of participants with the EducaDor program will be measured by the frequency rate in synchronous meetings; self-report of performance of proposed homework on a numerical scale from 0 to 10 during the intervention period; and by exercise adherence scale.
Maintenance of the intervention fidelity up to 6 months | up to 6 months
  The adherence of participants with the EducaDor program will be measured by the frequency rate in synchronous meetings; self-report of performance of proposed homework on a numerical scale from 0 to 10 during the intervention period; and by exercise adherence scale.
Assessment of the intervention penetration | through study completion, an average 24 months
  Penetration will be analyzed descriptively from the rate of public health users referred from each Primary Health Care unit.
Economic evaluation of the intervention | baseline; up to 6 months
  Economic evaluation will be analyzed from society perspective in a time horizon of 6 months (after the end of interventions and 6-month follow-up). The costs of intervention will be determined by maintenance and support technology costs, costs of monitoring data and staff, costs of training health professionals and project management, number and duration of phone calls and number of text messages sent to participants. The total costs of society will be estimated from the public and private health care costs, if possible (prescribed drugs, medical consultations, physical therapy care, visits to specialists, diagnostic exams, emergency services and hospitalization), patients costs (unprescribed drugs, complementary costs and transportation costs), and cmosts with loss of productivity (absenteeism and presenteeism) collected through a daily cost.
Assessment of the intervention sustainability | through study completion, an average 24 months
  Sustainability will be evaluated by a focus group interview with public health managers after presentation the results of the study to discuss the maintenance of the EducaDor program; and by response rate of synchronous group users and reasons for discontinuity the program through an individual qualitative interview

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Estadual do Centro-Oeste, Guarapuava, Paraná, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Baroni MP, Hespanhol L, Miyamoto GC, Daniel CR, Fernandes LG, Dos Reis FJJ, Pate JW, Saragiotto BT. Implementation of an online pain science education for chronic musculoskeletal pain in Brazilian public health system: protocol for a hybrid type III randomised controlled trial with economic evaluation. BMC Musculoskelet Disord. 2023 Apr 10;24(1):277. doi: 10.1186/s12891-023-06360-7. PMID 37038146